CLINICAL TRIAL: NCT00745563
Title: Testing the Effect of Intra-uterine Slow-Release Insemination (SRI) on the Pregnancy Rate in Women Designated for Artificial Insemination
Brief Title: Effects of Intra-uterine Slow-Release Insemination on Pregnancy Rate in Women Designated for Artificial Insemination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fertiligent (Industry)
Responsible Party: Dr. Hanna Levy, Fertiligent
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BRIDGE1 20/7/2008
Record Dates: First submitted 2008-08-30; First posted 2008-09-03 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2008-12

CONDITIONS: Infertility
Keywords: infertility; insemination; slow release
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Device: Fertiligent

INTERVENTIONS:
Device: Fertiligent — Fertility treatment by using the EVIE - Slow Release Insemination method

SUMMARY:
A couple that does not achieve pregnancy though regular attempts for a year are defined infertile couple. This condition is caused by faulty functioning of the reproduction system of the husband or wife or both. If there are no organic defects and there is no definite injury to the reproductive system (ova or spermatozoa), the specialist doctor generally decides to put the couple into a fertility treatment program. Artificial insemination is one of the important ways of achieving pregnancy.

Three common methods of artificial insemination:

1. Placement of a diaphragm that contains raw spermatozoa or isolated improved spermatozoa in an appropriate liquid solution (Cup insemination, CI) upon the cervix.
2. Spermatozoa injection (after improvement) through the vagina to the cervix (Intra-Cervical Insemination, ICI).
3. Spermatozoa injection (after improvement) directly into the uterus (IUI-Intra-Uterine Insemination).

The EVIE - Slow Release Insemination method:

The slow release insemination is utilizing a Grasby type MS16 pump for 3 hours. The release rate for motile spermatozoa is 50X103 per minute.

Advantages:

* Very close approximation of the natural procedure in which the spermatozoa arrive to the fertilization site over a long period.
* An extended "window of opportunities" for meeting between the ovum and spermatozoa will be longer.
* There is no loss of spermatozoa due to leaking as sometimes happens with single-time injection practiced in the IUI method.

Primary Endpoint:

Accumulation of 50 cycles of SRI- slow release insemination (study group) in addition to 50 cycles of regular IUI (control group). Two weeks after insemination Beta hCG test

Secondary Endpoints:

Four weeks after insemination - US Viability scan

Procedure:

Subjects will be women with fertility difficulties who are designated for IUI treatment. 100 insemination cycles will be conducted. (50 regular IUI and 50 EVIE-SRI). Subjects that were treated with the IUI method and who does not become pregnant will then be treated with the EVIE-Slow Release method and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary infertility designated for IUI treatment.
* Age of candidates: 20-40 years.
* Normal uterus x-ray.
* Women suffering from infertility on a background of non-ovulation.
* Infertility on a background of male problems (over 10 million of motile sperm cells per sample).
* Infertility on background of unexplained problem
* Same sex patients / single patient
* Written informed consent

Exclusion Criteria:

* Woman under the age of 20 or over the age of 40 years.
* Female infertility on mechanical background (different blockages, irregular uterus).
* Infertility on male background of medium to very low level of spermatozoa - less than 10 million motile sperm cells per sample.
* Men and women who are opposed to the random spermatozoa insemination method.
* Participants who are not willing to sign the Consent Form.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Accumulation of 50 cycles of SRI- slow release insemination (study group) in addition to 50 cycles of regular IUI (control group). Two weeks after insemination Beta hCG test | 2 weeks following procedure

SECONDARY OUTCOMES:
Four weeks after insemination - US Viability scan | 4 weeks following procedure

CONTACTS AND LOCATIONS:
Overall Officials: Martha Dirnfeld, Prof., Principal Investigator — Carmel medical Center, Haifa Israel
Locations (1):
- Carmel Medical Center, Haifa, Israel